CLINICAL TRIAL: NCT01550289
Title: Immunogenicity and Safety of a Tetravalent Dengue Vaccine in Healthy Adult Subjects Aged 18 to 45 Years in India.
Brief Title: Study of a Tetravalent Dengue Vaccine in Healthy Adult Subjects Aged 18 to 45 Years in India
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CYD47; UTN: U1111-1114-7909 (Other: WHO)
Record Dates: First submitted 2012-03-07; First posted 2012-03-09 (Estimated); Results first posted 2016-11-03 (Estimated); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Dengue; Dengue Fever; Dengue Hemorrhagic Fever
Keywords: Dengue Fever; Dengue Hemorrhagic Fever; CYD Dengue Vaccine; Dengue Virus; Flavivirus
MeSH Terms: conditions — Dengue; Severe Dengue | interventions — Solutions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1: CYD dengue vaccine (Experimental): Subjects will receive a dose of CYD dengue vaccine at 0, 6, and 12 months, respectively.
  Interventions: Biological: Live, attenuated, recombinant dengue serotype 1, 2, 3, 4 virus
- Group 2: Placebo (Placebo Comparator): Subjects will receive a dose of placebo at 0, 6, and 12 months, respectively
  Interventions: Biological: Placebo: NaCl 0.9% solution

INTERVENTIONS:
Biological: Live, attenuated, recombinant dengue serotype 1, 2, 3, 4 virus — 0.5 mL, Subcutaneous
  Other Names: CYD Dengue vaccine
  Arms: Group 1: CYD dengue vaccine
Biological: Placebo: NaCl 0.9% solution — 0.5 ml, Subcutaneous
  Arms: Group 2: Placebo

SUMMARY:
The aim of this study is to evaluate the immunogenicity and safety of the CYD dengue vaccine in India adult subjects.

Primary Objectives:

* To describe the neutralizing antibody response to each dengue virus serotype before the first vaccination and after each vaccination with CYD dengue vaccine in all subjects.
* To describe the safety of the CYD dengue vaccine after each dose in all subjects.

Secondary Objective:

* To detect symptomatic dengue cases occurring at any time in the trial.

DETAILED DESCRIPTION:
Participants will receive 3 doses of their randomized treatment (vaccine or placebo). Flavivirus status will be determined at baseline (before the first dose) and the vaccine immunogenicity assessment will be at 28 days after each vaccination. Reactogenicity data will be collected in all subjects after each dose. Serious adverse events and adverse events of special interest will be collected throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 45 years on the day of inclusion
* Informed consent form has been signed and dated by the subject (and by an independent witness, if applicable)
* Subject is able to attend all scheduled visits and to comply with all trial procedures
* Subject in good health, based on medical history and physical examination

Exclusion Criteria:

* Subject is pregnant, or lactating, or of childbearing potential (to be considered of non-childbearing potential, a female must be post-menopausal for at least 1 year, surgically sterile, or using an effective method of contraception or abstinence from at least 4 weeks prior to the first vaccination and until at least 4 weeks after the last vaccination)
* Participation in another clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 4 weeks preceding the first trial vaccination
* Planned participation in another clinical trial during the present trial period
* Planned receipt of any vaccine in the 4 weeks following any trial vaccination
* Receipt of blood or blood-derived products in the past 3 months, which might interfere with assessment of the immune response
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Known seropositivity for human immunodeficiency virus (HIV), hepatitis B, and hepatitis C reported by the subject
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine(s) used in the trial or to a vaccine containing any of the same substances
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion
* Current alcohol abuse or drug addiction that might interfere with the ability to comply with trial procedures
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Identified as an Investigator or employee of the Investigator or study center, with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 189 (Actual)
Dates: Start 2012-03; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur India Pvt Ltd
Locations (5):
- India (5):
  - Bangalore, Karnataka
  - Ludhiana, Punjab
  - Kolkata, West Bengal
  - New Delhi
  - Pune

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Result] Dubey AP, Agarkhedkar S, Chhatwal J, Narayan A, Ganguly S, Wartel TA, Bouckenooghe A, Menezes J. Immunogenicity and safety of a tetravalent dengue vaccine in healthy adults in India: A randomized, observer-blind, placebo-controlled phase II trial. Hum Vaccin Immunother. 2016;12(2):512-8. doi: 10.1080/21645515.2015.1076598. PMID 26291554
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 27 March 2012 to 28 June 2012 at 5 clinical centers in India.
Pre-assignment Details: A total of 189 participants who met all inclusion and no exclusion criteria were randomized and vaccinated in this trial; 187 were included in the Full Analysis Set.
Groups:
- CYD Dengue Vaccine Group: Healthy adult participants received 3 vaccinations of the CYD Dengue Vaccine.
- Placebo Group: Healthy adult participants received 3 vaccinations of placebo vaccine.
Period: Overall Study
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Started | 128 | 61
Completed | 115 | 57
Not Completed | 13 | 4
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 11 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CYD Dengue Vaccine Group | Placebo Group | Total
Number analyzed (Participants) | 126 | 61 | 187
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 126 | 61 | 187
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.5 (7.17) | 29.6 (6.41) | 29.5 (6.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 9 | 36
  Male | 99 | 52 | 151
Region of Enrollment [Count of Participants; unit: Participants]
  India | 126 | 61 | 187

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Antibody Titer ≥ 10 1/Dil Against Each Dengue Virus Serotype Before and After Each Vaccination With Either Tetravalent Dengue Vaccine or a Placebo
Description: Dengue neutralizing antibody levels were measured by dengue plaque reduction neutralization test (PRNT).
Time Frame: Pre-injection 1 and 28 days post each injection (up to 13 months post-injection 1)
Population: Dengue neutralizing antibody titers were assessed in the Full Analysis Set with available data for each time point.
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 126 | 61
Percentage of participants
  Serotype 1; Pre-injection 1 (N=126, 61) | 83.3 | 80.3
  Serotype 1; Post-injection 1 (N=125, 61) | 91.2 | 83.6
  Serotype 1; Post-injection 2 (N=117, 58) | 94.9 | 81.0
  Serotype 1; Post-injection 3 (N=115, 57) | 97.4 | 87.7
  Serotype 2; Pre-injection 1 (N=126, 61) | 83.3 | 86.9
  Serotype 2; Post-injection 1 (N=126, 61) | 94.4 | 88.5
  Serotype 2; Post-injection 2 (N=117, 58) | 99.1 | 84.5
  Serotype 2; Post-injection 3 (N=115, 57) | 97.4 | 91.2
  Serotype 3; Pre-injection 1 (N=126, 61) | 84.9 | 86.9
  Serotype 3; Post-injection 1 (N=126, 61) | 98.4 | 90.2
  Serotype 3; Post-injection 2 (N=117, 58) | 98.3 | 84.5
  Serotype 3; Post-injection 3 (N=115, 57) | 99.1 | 89.5
  Serotype 4; Pre-injection 1 (N=126, 61) | 77.0 | 80.3
  Serotype 4; Post-injection 1 (N=126, 61) | 96.0 | 85.2
  Serotype 4; Post-injection 2 (N=117, 57) | 99.1 | 78.9
  Serotype 4; Post-injection 3 (N=115, 57) | 100.0 | 84.2

2. Primary Outcome: Percentage of Participants With Antibody Titer ≥ 10 1/Dil Against at Least 1, 2, 3, or 4 Dengue Virus Serotypes Before and After Each Vaccination With Either Tetravalent Dengue Vaccine or a Placebo
Description: Dengue neutralizing antibody levels were measured by dengue plaque reduction neutralization test (PRNT).
Time Frame: Pre-injection 1 and 28 days post each injection (up to 13 months post-injection 1)
Population: Dengue neutralizing antibody titers were assessed in the Full Analysis Set with available data for each time point.
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 126 | 61
Percentage of participants
  At least 1 serotype; Pre-injection 1 (N=126, 61) | 86.5 | 88.5
  At least 1 serotype; Post-injection 1 (N=126, 61) | 99.2 | 90.2
  At least 1 serotype; Post-injection 2 (N=117, 58) | 100.0 | 86.2
  At least 1 serotype; Post-injection 3 (N=115, 57) | 100.0 | 91.2
  At least 2 serotypes; Pre-injection 1 (N=126, 61) | 84.1 | 85.2
  At least 2 serotypes; Post-injection 1 (N=126, 61) | 98.4 | 88.5
  At least 2 serotypes; Post-injection 2 (N=117, 58) | 98.3 | 82.8
  At least 2 serotypes; Post-injection 3 (N=115, 57) | 99.1 | 89.5
  At least 3 serotypes; Pre-injection 1 (N=126, 61) | 82.5 | 83.6
  At least 3 serotypes; Post-injection 1 (N=126, 61) | 92.1 | 88.5
  At least 3 serotypes; Post-injection 2 (N=117, 58) | 98.3 | 81.0
  At least 3 serotypes; Post-injection 3 (N=115, 57) | 97.4 | 87.7
  All 4 serotypes; Pre-injection 1 (N=126, 61) | 75.4 | 77.0
  All 4 serotypes; Post-injection 1 (N=126, 61) | 89.7 | 80.3
  All 4 serotypes; Post-injection 2 (N=117, 58) | 94.9 | 77.6
  All 4 serotypes; Post-injection 3 (N=115, 57) | 97.4 | 84.2

3. Primary Outcome: Summary of Geometric Mean Titers of Antibodies Against Each Dengue Serotype Before and After Each Vaccination With Either Tetravalent Dengue Vaccine or a Placebo
Description: Dengue neutralizing antibody levels were measured by dengue plaque reduction neutralization test (PRNT).
Time Frame: Pre-injection 1 and 28 days post each injection (up to 13 months post-injection 1)
Population: Geometric mean titers were assessed in the Full Analysis Set with available data for each time point.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilutions)
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 126 | 61
Titers (1/dilutions)
  Serotype 1; Pre-injection 1 (N=126, 61) | 184 [127 to 268] | 234 [133 to 409]
  Serotype 1; Post-injection 1 (N=125, 61) | 605 [410 to 892] | 288 [161 to 513]
  Serotype 1; Post-injection 2 (N=117, 58) | 556 [391 to 790] | 294 [159 to 543]
  Serotype 1; Post-injection 3 (N=115, 57) | 461 [340 to 625] | 268 [164 to 438]
  Serotype 2; Pre-injection 1 (N=126, 61) | 204 [141 to 294] | 243 [147 to 403]
  Serotype 2; Post-injection 1 (N=126, 61) | 720 [510 to 1015] | 300 [184 to 489]
  Serotype 2; Post-injection 2 (N=117, 58) | 787 [592 to 1045] | 288 [163 to 509]
  Serotype 2; Post-injection 3 (N=115, 57) | 484 [370 to 634] | 258 [163 to 410]
  Serotype 3; Pre-injection 1 (N=126, 61) | 219 [153 to 312] | 216 [131 to 354]
  Serotype 3; Post-injection 1 (N=126, 61) | 951 [691 to 1309] | 293 [180 to 478]
  Serotype 3; Post-injection 2 (N=117, 58) | 846 [635 to 1127] | 249 [143 to 434]
  Serotype 3; Post-injection 3 (N=115, 57) | 709 [552 to 911] | 268 [168 to 426]
  Serotype 4; Pre injection 1 (N=126, 61) | 55.4 [41.4 to 74.2] | 62.0 [42.0 to 91.5]
  Serotype 4; Post-injection 1 (N=126, 61) | 358 [271 to 472] | 78.7 [52.7 to 117]
  Serotype 4; Post-injection 2 (N=117, 57) | 289 [236 to 354] | 72.8 [46.6 to 114]
  Serotype 4; Post-injection 3 (N=115, 57) | 336 [271 to 417] | 91.9 [60.8 to 139]

4. Primary Outcome: Summary of Geometric Mean Titer Ratios of Antibodies Against Each Dengue Serotype Before and After Each Vaccination With Either Tetravalent Dengue Vaccine or a Placebo
Description: Dengue neutralizing antibody levels were measured by dengue plaque reduction neutralization test (PRNT).
Time Frame: Pre-injection 1 and 28 days post each injection (up to 13 months post-injection 1)
Population: Geometric mean titer ratios were assessed in the Full Analysis Set with available data for each time point.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer ratio
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 126 | 61
Titer ratio
  Serotype 1; Post-inj. 1/Pre-inj. 1 (N=125,61) | 3.23 [2.49 to 4.18] | 1.23 [1.02 to 1.49]
  Serotype 1; Post-inj. 2/Pre-inj. 1 (N=117,58) | 3.15 [2.46 to 4.04] | 1.26 [1.01 to 1.58]
  Serotype 1; Post-inj. 3/Pre-inj. 1 (N=115,57) | 2.64 [2.08 to 3.35] | 1.18 [0.838 to 1.66]
  Serotype 2; Post-inj. 1/Pre-inj. 1 (N=126,61) | 3.53 [2.76 to 4.52] | 1.23 [1.03 to 1.47]
  Serotype 2; Post-inj. 2/Pre-inj. 1 (N=117,58) | 3.83 [2.84 to 5.18] | 1.17 [0.951 to 1.45]
  Serotype 2; Post-inj. 3/Pre-inj. 1 (N=115,57) | 2.38 [1.81 to 3.11] | 1.05 [0.791 to 1.41]
  Serotype 3; Post-inj. 1/Pre-inj. 1 (N=126,61) | 4.35 [3.34 to 5.68] | 1.36 [1.09 to 1.69]
  Serotype 3; Post-inj. 2/Pre-inj. 1 (N=117,58) | 3.97 [2.99 to 5.28] | 1.13 [0.888 to 1.44]
  Serotype 3; Post-inj. 3/Pre-inj. 1 (N=115,57) | 3.39 [2.61 to 4.40] | 1.22 [0.869 to 1.72]
  Serotype 4; Post-inj. 1/Pre-inj. 1 (N=126,61) | 6.46 [4.74 to 8.79] | 1.27 [1.00 to 1.61]
  Serotype 4; Post-inj. 2/Pre-inj. 1 (N=117,57) | 5.16 [3.98 to 6.68] | 1.15 [0.920 to 1.45]
  Serotype 4; Post-inj. 3/Pre-inj. 1 (N=115,57) | 6.11 [4.81 to 7.77] | 1.44 [1.09 to 1.90]

5. Primary Outcome: Percentage of Participants With Solicited Injection-site and Systemic Reactions After Any and Each Injection With Either CYD Dengue Tetravalent Vaccine or a Placebo
Description: Solicited injection-site: Pain, Erythema, and Swelling. Solicited systemic reactions: Fever (Temperature), Headache, Malaise, Myalgia, and Asthenia. Grade 3 Solicited Injection site reactions: Pain Significant; prevents daily activities; Erythema and Swelling >100 mm. Grade 3 Solicited systemic reactions: Fever ≥39.0˚C; Headache, Malaise, Myalgia, and Asthenia Significant; prevents daily activities.
Time Frame: Day 0 up to Day 14 post each injection
Population: Solicited injection-site and systemic reactions were assessed in the Safety Analysis Set with available data for each time point.
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 127 | 61
Percentage of participants
  Injection-site Pain; Post-Any inj. (N=126, 61) | 9.5 | 4.9
  Grade 3 Inj.-site Pain; Post-Any inj. (N=126, 61) | 0.0 | 0.0
  Injection-site Erythema; Post-Any inj. (N=126, 61) | 0.0 | 0.0
  Grade 3 Inj.-site Erythema;Post-Any inj (N=126,61) | 0.0 | 0.0
  Injection-site Swelling; Post-Any inj. (N=126, 61) | 0.0 | 0.0
  Grade 3 Inj.-site Swelling;PostAny inj (N=126,61) | 0.0 | 0.0
  Injection-site Pain; Post-inj. 1 (N=126, 61) | 6.3 | 4.9
  Grade 3 Inj.-site Pain; Post-inj. 1 (N=126, 61) | 0.0 | 0.0
  Injection-site Erythema; Post-inj. 1 (N=126, 61) | 0.0 | 0.0
  Grade 3 Inj.-site Erythema; Post-inj 1 (N=126,61) | 0.0 | 0.0
  Injection-site Swelling; Post-inj. 1 (N=126, 61) | 0.0 | 0.0
  Grade 3 Inj.-site Swelling; Post-inj. 1 (N=126,61) | 0.0 | 0.0
  Injection-site Pain; Post-inj. 2 (N=117, 58) | 1.7 | 3.4
  Grade 3 Inj.-site Pain; Post-inj. 2 (N=117, 58) | 0.0 | 0.0
  Injection-site Erythema; Post-inj. 2 (N=117, 58) | 0.0 | 0.0
  Grade 3 Inj.-site Erythema; Post-inj 2 (N=117,58) | 0.0 | 0.0
  Injection-site Swelling; Post-inj. 2 (N=117, 58) | 0.0 | 0.0
  Grade 3 Inj.-site Swelling; Post-inj. 2 (N=117,58) | 0.0 | 0.0
  Injection-site Pain; Post-inj. 3 (N=115, 57) | 2.6 | 0.0
  Grade 3 Inj.-site Pain; Post-inj. 3 (N=115, 57) | 0.0 | 0.0
  Injection-site Erythema; Post-inj. 3 (N=115, 57) | 0.0 | 0.0
  Grade 3 Inj.-site Erythema; Post-inj 3 (N=115,57) | 0.0 | 0.0
  Injection-site Swelling; Post-inj. 3 (N=115, 57) | 0.0 | 0.0
  Grade 3 Inj.-site Swelling; Post-inj. 3 (N=115,57) | 0.0 | 0.0
  Fever; Post-Any inj. (N=126, 61) | 5.6 | 1.6
  Grade 3 Fever; Post-Any inj. (N=126, 61) | 0.8 | 0.0
  Headache; Post Any-inj. (N=126, 61) | 7.9 | 4.9
  Grade 3 Headache; Post-Any inj. (N=126, 61) | 1.6 | 1.6
  Malaise; Post-Any inj. (N=126, 61) | 8.7 | 4.9
  Grade 3 Malaise; Post-Any inj. (N=126, 61) | 0.8 | 0.0
  Myalgia; Post Any inj. (N=126, 61) | 9.5 | 4.9
  Grade 3 Myalgia; Post-Any inj. (N=126, 61) | 0.0 | 1.6
  Asthenia; Post-Any inj. (N=126, 61) | 11.1 | 4.9
  Grade 3 Asthenia; Post-Any inj. (N=126, 61) | 0.8 | 0.0
  Fever; Post-inj. 1 (N=125, 60) | 4.8 | 0.0
  Grade 3 Fever; Post-inj. 1 (N=125, 60) | 0.8 | 0.0
  Headache; Post-inj. 1 (N=126, 61) | 5.6 | 4.9
  Grade 3 Headache; Post-inj. 1 (N=126, 61) | 1.6 | 1.6
  Malaise; Post-inj. 1 (N=126, 61) | 7.1 | 4.9
  Grade 3 Malaise; Post-inj. 1 (N=126, 61) | 0.0 | 0.0
  Myalgia; Post-inj. 1 (N=126, 61) | 7.9 | 4.9
  Grade 3 Myalgia; Post inj. 1 (N=126, 61) | 0 | 1.6
  Asthenia; Post-inj. 1 (N=126, 61) | 9.5 | 4.9
  Grade 3 Asthenia; Post inj. 1 (N=126, 61) | 0.0 | 0.0
  Fever; Post-inj. 2 (N=117, 58) | 0.9 | 1.7
  Grade 3 Fever; Post-inj. 2 (N=117, 58) | 0.0 | 0.0
  Headache; Post-inj. 2 (N=117, 58) | 1.7 | 0.0
  Grade 3 Headache; Post-inj. 2 (N=117, 58) | 0.0 | 0.0
  Malaise; Post-inj. 2 (N=117, 58) | 0.9 | 0.0
  Grade 3 Malaise; Post-inj. 2 (N=117, 58) | 0.9 | 0.0
  Myalgia; Post-inj. 2 (N=117, 58) | 1.7 | 0.0
  Grade 3 Myalgia; Post-inj. 2 (N=117, 58) | 0.0 | 0.0
  Asthenia; Post-inj. 2 (N=117, 58) | 2.6 | 0.0
  Grade 3 Asthenia; Post-inj. 2 (N=117, 58) | 0.9 | 0.0
  Fever; Post-inj. 3 (N=113, 57) | 0.0 | 0.0
  Grade 3 Fever; Post inj. 3 (N=113, 57) | 0.0 | 0.0
  Headache; Post-inj. 3 (N=115, 57) | 0.9 | 0.0
  Grade 3 Headache; Post-inj. 3 (N=115, 57) | 0.0 | 0.0
  Malaise; Post-inj. 3 (N=115, 57) | 0.9 | 0.0
  Grade 3 Malaise; Post-inj. 3 (N=115, 57) | 0.0 | 0.0
  Myalgia; Post-inj. 3 (N=115, 57) | 0.0 | 0.0
  Grade 3 Myalgia; Post-inj. 3 (N=115, 57) | 0.0 | 0.0
  Asthenia; Post-inj. 3 (N=115, 57) | 0.0 | 0.0
  Grade 3 Asthenia; Post-inj. 3 (N=115, 57) | 0.0 | 0.0

6. Secondary Outcome: Percentage of Flavivirus-Immune Participants With Antibody Titer ≥ 10 1/Dil Against Each Dengue Serotype Before and After Each Tetravalent Dengue Vaccine or a Placebo
Description: Dengue neutralizing antibody levels were measured by dengue plaque reduction neutralization test (PRNT). Flavivirus (FV) immune participants at baseline are defined as those participants with ≥10 (1/dil) for at least one serotype with the parental dengue virus strain or for Japanese encephalitis (JE) virus.
Time Frame: Pre-injection 1 and 28 days post each injection (up to 13 months post-injection 1)
Population: Dengue neutralizing antibody titers were assessed in the Full Analysis Set with available data for each time point.
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 113 | 56
Percentage of participants
  Serotype 1; Pre-injection 1 (N=113, 56) | 92.9 | 87.5
  Serotype 1; Post-injection 1 (N=112, 56) | 96.4 | 89.3
  Serotype 1; Post-injection 2 (N=104, 53) | 99.0 | 88.7
  Serotype 1; Post-injection 3 (N=102, 52) | 100.0 | 94.2
  Serotype 2; Pre-injection 1 (N=113, 56) | 92.9 | 94.6
  Serotype 2; Post-injection 1 (N=113, 56) | 98.2 | 94.6
  Serotype 2; Post-injection 2 (N=104, 53) | 100.0 | 92.5
  Serotype 2; Post-injection 3 (N=102, 52) | 100.0 | 98.1
  Serotype 3; Pre-injection 1 (N=113, 56) | 94.7 | 94.6
  Serotype 3; Post-injection 1 (N=113, 56) | 100.0 | 96.4
  Serotype 3; Post-injection 2 (N=104, 53) | 100.0 | 92.5
  Serotype 3; Post-injection 3 (N=102, 52) | 100.0 | 96.2
  Serotype 4; Pre-injection 1 (N=113, 56) | 85.8 | 87.5
  Serotype 4; Post-injection 1 (N=113, 56) | 98.2 | 91.1
  Serotype 4; Post-injection 2 (N=104, 52) | 100.0 | 86.5
  Serotype 4; Post-injection 3 (N=102, 52) | 100.0 | 90.4

7. Secondary Outcome: Percentage of Flavivirus-non Immune Participants With Antibody Titer < 10 1/Dil Against Each Dengue Serotype Before and After Each Tetravalent Dengue Vaccine or a Placebo
Description: Dengue neutralizing antibody levels were measured by dengue plaque reduction neutralization test (PRNT). Flavivirus (FV) non-immune participants at baseline are defined as those participants with <10 (1/dil) for all serotypes with parental dengue virus strains and for Japanese encephalitis (JE) virus.
Time Frame: Pre-injection 1 and 28 days post each injection (up to 13 months post-injection 1)
Population: Dengue neutralizing antibody titers were assessed in the Full Analysis Set with available data for each time point.
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 13 | 5
Percentage of participants
  Serotype 1; Pre-injection 1 (N=13, 5) | 0.0 | 0.0
  Serotype 1; Post-injection 1 (N=13, 5) | 46.2 | 20.0
  Serotype 1; Post-injection 2 (N=13, 5) | 61.5 | 0.0
  Serotype 1; Post-injection 3 (N=13, 5) | 76.9 | 20.0
  Serotype 2; Pre-injection 1 (N=13, 5) | 0.0 | 0.0
  Serotype 2; Post-injection 1 (N=13, 5) | 61.5 | 20.0
  Serotype 2; Post-injection 2 (N=13, 5) | 92.3 | 0.0
  Serotype 2; Post injection 3 (N=13, 5) | 76.9 | 20.0
  Serotype 3; Pre-injection 1 (N=13, 5) | 0.0 | 0.0
  Serotype 3; Post-injection 1 (N=13, 5) | 84.6 | 20.0
  Serotype 3; Post-injection 2 (N=13, 5) | 84.6 | 0.0
  Serotype 3; Post-injection 3 (N=13, 5) | 92.3 | 20.0
  Serotype 4; Pre-injection 1 (N=13, 5) | 0.0 | 0.0
  Serotype 4; Post-injection 1 (N=13, 5) | 76.9 | 20.0
  Serotype 4; Post-injection 2 (N=13, 5) | 92.3 | 0.0
  Serotype 4; Post-injection 3 (N=13, 5) | 100.0 | 20.0

8. Secondary Outcome: Percentage of Flavivirus-Immune Participants With Antibody Titer ≥ 10 1/Dil Against at Least 1, 2, 3, or 4 Dengue Serotypes Before and After Each Tetravalent Dengue Vaccine or a Placebo
Description: as for outcome 6
Time Frame: Pre-injection 1 and 28 days post each injection (up to 13 months post-injection 1)
Population: Dengue neutralizing antibody titers were assessed in the Full Analysis Set with available data for each time point.
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 113 | 56
Percentage of participants
  At least 1 serotype; Pre-injection 1 (N=113, 56) | 96.5 | 96.4
  At least 1 serotype; Post-injection 1 (N=113, 56) | 100.0 | 96.4
  At least 1 serotype; Post-injection 2 (N=104, 53) | 100.0 | 94.3
  At least 1 serotype; Post-injection 3 (N=102, 52) | 100.0 | 98.1
  At least 2 serotypes; Pre-injection 1 (N=113, 56) | 93.8 | 92.9
  At least 2 serotypes; Post-injection 1 (N=113, 56) | 100.0 | 94.6
  At least 2 serotypes; Post-injection 2 (N=104, 53) | 100.0 | 90.6
  At least 2 serotypes; Post-injection 3 (N=102, 52) | 100.0 | 96.2
  At least 3 serotypes; Pre-injection 1 (N=113, 56) | 92.0 | 91.1
  At least 3 serotypes; Post-injection 1 (N=113, 56) | 96.5 | 94.6
  At least 3 serotypes; Post-injection 2 (N=104, 53) | 100.0 | 88.7
  At least 3 serotypes; Post-injection 3 (N=102, 52) | 100.0 | 94.2
  All 4 serotypes; Pre-injection 1 (N=113, 56) | 84.1 | 83.9
  All 4 serotypes; Post-injection 1 (N=113, 56) | 95.6 | 85.7
  All 4 serotypes; Post-injection 2 (N=104, 53) | 99.0 | 84.9
  All 4 serotypes; Post-injection 3 (N=102, 52) | 100.0 | 90.4

9. Secondary Outcome: Percentage of Flavivirus-non Immune Participants With Antibody Titer < 10 1/Dil Against at Least 1, 2, 3, or 4 Dengue Serotypes Before and After Each Tetravalent Dengue Vaccine or a Placebo
Description: Dengue neutralizing antibody levels were measured by dengue plaque reduction neutralization test (PRNT). Flavivirus (FV) non immune participants at baseline are defined as those participants with <10 (1/dil) for all serotypes with parental dengue virus strains and for Japanese encephalitis (JE) virus.
Time Frame: Pre-injection 1 and 28 days post each injection (up to 13 months post-injection 1)
Population: Dengue neutralizing antibody titers were assessed in the Full Analysis Set with available data for each time point.
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 13 | 5
Percentage of participants
  At least 1 serotype; Pre-injection 1 (N=13, 5) | 0.0 | 0.0
  At least 1 serotype; Post-injection 1 (N=13, 5) | 92.3 | 20.0
  At least 1 serotype; Post-injection 2 (N=13, 5) | 100.0 | 0.0
  At least 1 serotype; Post-injection 3 (N=13, 5) | 100.0 | 20.0
  At least 2 serotypes; Pre-injection 1 (N=13, 5) | 0.0 | 0.0
  At least 2 serotypes; Post-injection 1 (N=13, 5) | 84.6 | 20.0
  At least 2 serotypes; Post-injection 2 (N=13, 5) | 84.6 | 0.0
  At least 2 serotypes; Post-injection 3 (N=13, 5) | 92.3 | 20.0
  At least 3 serotypes; Pre-injection 1 (N=13, 5) | 0.0 | 0.0
  At least 3 serotypes; Post-injection 1 (N=13, 5) | 53.8 | 20.0
  At least 3 serotypes; Post-injection 2 (N=13, 5) | 84.6 | 0.0
  At least 3 serotypes; Post-injection 3 (N=13, 5) | 76.9 | 20.0
  All 4 serotypes; Pre-injection 1 (N=13, 5) | 0.0 | 0.0
  All 4 serotypes; Post-injection 1 (N=13, 5) | 38.5 | 20.0
  All 4 serotypes; Post-injection 2 (N=13, 5) | 61.5 | 0.0
  All 4 serotypes; Post-injection 3 (N=13, 5) | 76.9 | 20.0

10. Secondary Outcome: Summary of Geometric Mean Titers of Antibodies Against Each Dengue Serotype In Flavivirus-Immune Participants Before and After Each Vaccination With Either Tetravalent Dengue Vaccine or a Placebo
Description: as for outcome 6
Time Frame: Pre-injection 1 and 28 days post each injection (up to 13 months post-injection 1)
Population: Geometric mean titers were assessed in the Full Analysis Set with available data for each time point.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilutions)
Groups:
- CYD Dengue Vaccine Group: Healthy adult participants who received 3 vaccinations of the CYD Dengue Vaccine.
- Placebo Group: Healthy adult participants who received 3 vaccinations of placebo vaccine.
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 113 | 56
Titers (1/dilutions)
  Serotype 1; Pre-injection 1 (N=113, 56) | 279 [199 to 392] | 329 [196 to 553]
  Serotype 1; Post-injection 1 (N=112, 56) | 925 [656 to 1304] | 401 [232 to 691]
  Serotype 1; Post-injection 2 (N=104, 53) | 807 [591 to 1101] | 432 [245 to 760]
  Serotype 1; Post-injection 3 (N=102, 52) | 636 [485 to 834] | 362 [235 to 558]
  Serotype 2; Pre-injection 1 (N=113, 56) | 312 [225 to 432] | 344 [221 to 537]
  Serotype 2; Post-injection 1 (N=113, 56) | 1030 [765 to 1385] | 413 [268 to 636]
  Serotype 2; Post-injection 2 (N=104, 53) | 1010 [792 to 1288] | 422 [254 to 702]
  Serotype 2; Post-injection 3 (N=102, 52) | 624 [493 to 790] | 357 [242 to 528]
  Serotype 3; Pre-injection 1 (N=113, 56) | 338 [249 to 458] | 302 [195 to 469]
  Serotype 3; Post-injection 1 (N=113, 56) | 1324 [1002 to 1749] | 405 [263 to 623]
  Serotype 3; Post-injection 2 (N=104, 53) | 1131 [879 to 1455] | 361 [219 to 594]
  Serotype 3; Post-injection 3 (N=102, 52) | 912 [726 to 1145] | 368 [248 to 547]
  Serotype 4; Pre-injection 1 (N=113, 56) | 73.1 [55.1 to 96.9] | 77.6 [53.6 to 112]
  Serotype 4; Post-injection 1 (N=113, 56) | 424 [325 to 554] | 99.1 [67.8 to 145]
  Serotype 4; Post-injection 2 (N=104, 52) | 346 [287 to 417] | 94.2 [61.6 to 144]
  Serotype 4; Post-injection 3 (N=102, 52) | 387 [309 to 485] | 117 [79.7 to 172]

11. Secondary Outcome: Summary of Geometric Mean Titer Ratios of Antibodies Against Each Dengue Serotype In Flavivirus-Immune Participants Before and After Each Vaccination With Either Tetravalent Dengue Vaccine or a Placebo
Description: as for outcome 6
Time Frame: Pre-injection 1 and 28 days post each injection (up to 13 months post-injection 1)
Population: Geometric mean titers ratios were assessed in the Full Analysis Set with available data for each time point.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer ratio
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 113 | 56
Titer ratio
  Serotype 1; Post-inj. 1/Pre-inj. 1 (N=112,56) | 3.24 [2.47 to 4.25] | 1.22 [0.994 to 1.49]
  Serotype 1; Post-inj. 2/Pre-inj. 1 (N=104,53) | 2.93 [2.28 to 3.77] | 1.29 [1.01 to 1.65]
  Serotype 1; Post-inj. 3/Pre-inj. 1 (N=102,52) | 2.31 [1.82 to 2.94] | 1.10 [0.786 to 1.55]
  Serotype 2; Post-inj. 1/Pre-inj. 1 (N=113,56) | 3.30 [2.59 to 4.20] | 1.20 [1.01 to 1.43]
  Serotype 2; Post-inj. 2/Pre-inj. 1 (N=104,53) | 3.09 [2.34 to 4.08] | 1.19 [0.946 to 1.50]
  Serotype 2; Post-inj. 3/Pre-inj. 1 (N=102,52) | 1.91 [1.49 to 2.45] | 1.00 [0.746 to 1.35]
  Serotype 3; Post-inj. 1/Pre-inj. 1 (N=113,56) | 3.92 [3.00 to 5.13] | 1.34 [1.07 to 1.69]
  Serotype 3; Post-inj. 2/Pre-inj. 1 (N=104,53) | 3.32 [2.50 to 4.41] | 1.15 [0.878 to 1.50]
  Serotype 3; Post-inj. 3/Pre-inj. 1 (N=102,52) | 2.71 [2.10 to 3.49] | 1.17 [0.820 to 1.67]
  Serotype 4; Post-inj. 1/Pre-inj. 1 (N=113,56) | 5.80 [4.23 to 7.96] | 1.28 [0.988 to 1.65]
  Serotype 4; Post-inj. 2/Pre-inj. 1 (N=104,52) | 4.86 [3.48 to 5.99] | 1.17 [0.912 to 1.50]
  Serotype 4; Post-inj. 3/Pre-inj. 1 (N=102,52) | 5.18 [4.03 to 6.66] | 1.43 [1.06 to 1.93]

12. Secondary Outcome: Summary of Geometric Mean Titers of Antibodies Against Each Dengue Serotype In Flavivirus Non-immune Participants Before and After Each Vaccination With Either Tetravalent Dengue Vaccine or a Placebo
Description: as for outcome 9
Time Frame: Pre-injection 1 and 28 days post each injection (up to 13 months post-injection 1)
Population: Geometric mean titers were assessed in the Full Analysis Set with available data for each time point.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilutions)
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 13 | 5
Titers (1/dilutions)
  Serotype 1; Pre-injection 1 (N=13, 5) | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00]
  Serotype 1; Post-injection 1 (N=13, 5) | 15.5 [5.83 to 41.3] | 7.01 [2.75 to 17.9]
  Serotype 1; Post-injection 2 (N=13, 5) | 28.2 [9.88 to 80.4] | 5.00 [5.00 to 5.00]
  Serotype 1; Post-injection 3 (N=13, 5) | 37.1 [16.0 to 86.5] | 11.8 [1.09 to 126]
  Serotype 2; Pre-injection 1 (N=13, 5) | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00]
  Serotype 2; Post-injection 1 (N=13, 5) | 32.1 [9.14 to 112] | 8.27 [2.04 to 33.5]
  Serotype 2; Post-injection 2 (N=13, 5) | 107 [27.9 to 410] | 5.00 [5.00 to 5.00]
  Serotype 2; Post-injection 3 (N=13, 5) | 66.8 [22.8 to 196] | 8.93 [1.78 to 44.7]
  Serotype 3; Pre-injection 1 (N=13, 5) | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00]
  Serotype 3; Post-injection 1 (N=13, 5) | 53.8 [17.7 to 163] | 5.96 [3.66 to 9.69]
  Serotype 3; Post-injection 2 (N=13, 5) | 83.1 [30.3 to 228] | 5.00 [5.00 to 5.00]
  Serotype 3; Post-injection 3 (N=13, 5) | 98.6 [48.1 to 202] | 9.72 [1.53 to 61.6]
  Serotype 4; Pre-injection 1 (N=13, 5) | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00]
  Serotype 4; Post-injection 1 (N=13, 5) | 81.8 [25.0 to 267] | 5.96 [3.66 to 9.69]
  Serotype 4; Post-injection 2 (N=13, 5) | 68.4 [33.3 to 141] | 5.00 [5.00 to 5.00]
  Serotype 4; Post-injection 3 (N=13, 5) | 111 [79.9 to 155] | 7.29 [2.56 to 20.8]

13. Secondary Outcome: Summary of Geometric Mean Titer Ratios of Antibodies Against Each Dengue Serotype In Flavivirus Non-immune Participants Before and After Each Vaccination With Either Tetravalent Dengue Vaccine or a Placebo
Description: as for outcome 6
Time Frame: Pre-injection 1 and 28 days post each injection (up to 13 months post-injection 1)
Population: Geometric mean titers ratios were assessed in the Full Analysis Set with available data for each time point.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer ratio
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 13 | 5
Titer ratio
  Serotype 1; Post-inj. 1/Pre-inj. 1 (N=13,5) | 3.10 [1.17 to 8.25] | 1.40 [0.549 to 3.57]
  Serotype 1; Post-inj. 2/Pre-inj. 1 (N=13,5) | 5.64 [1.98 to 16.1] | 1.00 [1.00 to 1.00]
  Serotype 1; Post-inj. 3/Pre-inj. 1 (N=13,5) | 7.43 [3.19 to 17.3] | 2.35 [0.219 to 25.3]
  Serotype 2; Post-inj. 1/Pre-inj. 1 (N=13,5) | 6.41 [1.83 to 22.5] | 1.65 [0.409 to 6.70]
  Serotype 2; Post-inj. 2/Pre-inj. 1 (N=13,5) | 21.4 [5.59 to 81.9] | 1.00 [1.00 to 1.00]
  Serotype 2; Post-inj. 3/Pre-inj. 1 (N=13,5) | 13.4 [4.56 to 39.1] | 1.79 [0.357 to 8.95]
  Serotype 3; Post-inj. 1/Pre-inj. 1 (N=13,5) | 10.8 [3.55 to 32.6] | 1.58 [0.441 to 5.69]
  Serotype 3; Post-inj. 2/Pre-inj. 1 (N=13,5) | 16.6 [6.06 to 45.5] | 1.00 [1.00 to 1.00]
  Serotype 3; Post-inj. 3/Pre-inj. 1 (N=13,5) | 19.7 [9.63 to 40.4] | 1.94 [0.307 to 12.3]
  Serotype 4; Post-inj. 1/Pre-inj. 1 (N=13,5) | 16.4 [5.01 to 53.4] | 1.19 [0.733 to 1.94]
  Serotype 4; Post-inj. 2/Pre-inj. 1 (N=13,5) | 13.7 [6.66 to 28.1] | 1.00 [1.00 to 1.00]
  Serotype 4; Post-inj. 3/Pre-inj. 1 (N=13,5) | 22.2 [16.0 to 31.0] | 1.46 [0.511 to 4.16]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Day 0 up to 1 year post injection 1.
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 1/127 | 1/61
Other Adverse Events (participants affected / at risk) | 14/127 | 3/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CYD Dengue Vaccine Group (N=127) | Placebo Group (N=61)
Anaemia megaloblastic (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | CYD Dengue Vaccine Group (N=127) | Placebo Group (N=61)
Injection site Pain (General disorders) | 12 (12) | 3 (3)
Fever (General disorders) | 7/126 (7) | 1 (1)
Headache (Nervous system disorders) | 10/126 (10) | 3 (3)
Malaise (General disorders) | 11/126 (11) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 12/126 (12) | 3 (3)
Asthenia (General disorders) | 14/126 (14) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.